CLINICAL TRIAL: NCT01689389
Title: Description of the Use of Quetiapine Extended Release (XR) in Real-life Practice in France
Brief Title: Description of the Use of Quetiapine Extended Release (XR) in Real-life Practice in France. An Observational Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NFR-SER-2012/1
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia; Bipolar Episodes
Keywords: Schizophrenia; Bipolar episodes; France; Xeroquel; Real-life
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Main study population: All eligible patients receiving Quetiapine XR for the first time in the inclusion period regardless the diagnosed disease or the patients' age.
  Patients aged 18 years and over and diagnosed with bipolar disorder or schizophrenia according to DSM-IV criteria will be followed during 12 months.
- Schizophrenia SoC sample: Patients would have to be prescribed for the first time with a new (not used during the preceding 3 months) atypical antipsychotic other than Quetiapine XR (irrespective this new atypical antipsychotic is preceded or not by another atypical antipsychotic).
- Bipolar SoC sample: Patients would have to be prescribed a new (not used during the preceding 3 months) antidepressant [N06A], antipsychotic (other than Quetiapine XR) [N05A] or mood stabilizer (including lithium [N05AN], valproate [N03AG01], and lamotrigine [N03AX09].

SUMMARY:
The aim of the study is to describe patient characteristics (demographic and clinical) and the patterns of use of Quetiapine XR in patients receiving the drug for the first time in real-life practice regardless the final diagnosis.

DETAILED DESCRIPTION:
Description of the use of Quetiapine Extended Release (XR) in real-life practice in France

ELIGIBILITY:
Inclusion Criteria:

* New patients treated with Xeroquel XR
* Patients aged 18 years and over
* Diagnosis of bipolar disorder or schizophrenia according to DSM-IV criteria

Exclusion Criteria:

* Patient included in a therapeutic trial (Huriet-Serusclat Act)
* Patient refusing to participate in the study
* Pregnant women

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital, clinic
Sampling Method: Probability Sample
Enrollment: 2292 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of variables related with how the drug is prescribed and used by the patient. | At inclusion
  Variables related with how the drug is prescribed and used by the patient [doses in mg/day, titration (yes/no), time of administration (morning/middle of the day/afternoon/evening), concomitant treatments] are going to be described.
Description of patient's socio-demographics profile. | At inclusion
  Age, gender, educational and professional status, co-habitation are going to be described.
Descriptive analysis of medical history. | At inclusion
  Diagnosis, family history of psychiatric disorders, number of suicidal attempts within the last 12 months, co-morbidities, treatments received during the last 12 months, laboratory and exam data will be included in the description.
Severity of the disease measured by Clinical Global Impressions Scale - Severity (CGI-S). | At inclusion
  The Clinical Global Impressions Scale - Severity (CGI-S) assesses the clinician's impression of the current state of the patient's illness.
  The following scores can be given: 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill patients.

SECONDARY OUTCOMES:
Change in Clinical Global Impressions Scale - Severity (CGI-S) during the treatment. | From baseline to 12 months
  The Clinical Global Impressions Scale - Severity (CGI-S) assesses the clinician's impression of the current state of the patient's illness.
  The following scores can be given: 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill patients.
Quetiapine XR and concomitant treatment stop, stop date, reasons to stop, restart, restart date, reasons to restart. | From baseline to 12 months
Descriptive analysis of the treatment changes: drug switches. | From baseline to 12 months
Description of patterns of healthcare management resource use related with psychiatric disorders under investigation. | From baseline to 12 months
Change in Body Mass Index (BMI). | From baseline to 12 months
Laboratory tests- cholesterol. | From baseline to 12 months
  Blood test- cholesterol.
Descriptive analysis of all adverse events. | From baseline to 12 months
Relapses (only for the schizophrenia subpopulation). | From baseline to 12 months
  New psychiatric hospitalisation, deterioration of the CGI-S (Clinical Global Impressions Scale - Severity) by at least 3 points for a baseline score of 1, at least 2 points for a baseline score of 2 or 3, at least 1 point for a baseline score of 4.
Laboratory tests- glycemia. | From baseline to 12 months
  Blood test- glycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FALISSARD, Pr, Principal Investigator — Paris; Pierre-Michel LLORCA, Pr, Principal Investigator — Clermont-Ferrand
Locations (19):
- France (19):
  - Research Site, Argenteuil
  - Research Site, Belley
  - Research Site, Castelmaurou
  - Reserach Site, Cavaillon
  - Research Site, Les Mureaux
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nîmes
  - Research SIte, Obernai
  - Research Site, Paris
  - Research Site, Rennes
  - research Site, Saint-Dizier
  - Research Site, Saint-Égrève
  - Research Site, Saintes
  - Research Site, Sens
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Ussel

REFERENCES:
- See also: NIS-NFR-SER-2012/1 SUMMARY SYNOPSIS — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=928&filename=NIS-NFR-SER-2012-1_SUMMARY_SYNOPSIS.pdf